CLINICAL TRIAL: NCT02871817
Title: The Correlation of the Checkup Vision Assessment System to Standard In Office Visual Assessment
Brief Title: A Comparison of the Checkup Vision Assessment System to Standard Vision Assessment Tools
Acronym: CLEAR
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Digisight Technologies, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: SPD02000-01
Record Dates: First submitted 2016-07-18; First posted 2016-08-18 (Estimated); Last update posted 2018-01-26 (Actual); Status verified 2018-01

CONDITIONS: Age - Related Macular Degeneration; Diabetic Retinopathy; Metamorphopsia
Keywords: Near Corrected Visual Acuity; Early Treatment Diabetes Retinopathy Study; Amsler Grid; Home Monitoring
MeSH Terms: conditions — Macular Degeneration; Diabetic Retinopathy; Vision Disorders

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- Normal Vision: Patients without significant vision deficit (20/20 vision), when eligible and providing informed consent, assigned to evaluation with Paxos Checkup Study Mobile Medical Application
  Interventions: Other: Paxos Checkup Study Mobile Medical Application
- Age-related macular degeneration: Patients presenting with dry AMD or neovascular (wet) AMD, when eligible and providing informed consent, assigned to evaluation with Paxos Checkup Study Mobile Medical Application
  Interventions: Other: Paxos Checkup Study Mobile Medical Application
- Diabetic retinopathy: Patients presenting with Diabetic Retinopathy, when eligible and providing informed consent, assigned to evaluation with Paxos Checkup Study Mobile Medical Application
  Interventions: Other: Paxos Checkup Study Mobile Medical Application

INTERVENTIONS:
Other: Paxos Checkup Study Mobile Medical Application — The Digisight Paxos Checkup TM is mobile vision assessment system which consists of an application installed on a mobile device with an Internet connection, an Internet Cloud-based vision care network and a web site. The Paxos Checkup app contains a set of quantitative near vision tests, which a patient can take at home or elsewhere using an Internet capable mobile device.
  Other Names: Checkup Study

SUMMARY:
The CLEAR study is testing the level of agreement between visual acuity and Amsler grid testing using a mobile vision testing application, Checkup Study, and standard in office methods. In addition the percent of patients able to successfully complete home testing on the digital device will be assessed.

DETAILED DESCRIPTION:
BACKGROUND AND INTRODUCTION Neovascular Age - related Macular Degeneration (AMD) is the most common cause of vision loss in subjects over the age of 60. Today in the US over 15 million people live with some form of AMD, and approximately 1.6-1.75 million people have neovascular AMD associated with vision loss. Approximately 200,000 new cases are diagnosed in the US annually; worldwide, approximately 500,000 new cases are diagnosed each year. With the aging of the overall population, prevalence of all forms of AMD is expected to rise to as many as 42 million by 2030, and it is projected that as many as 8 million seniors are at risk for losing vision from AMD within the next 5 years. Economic analysis indicates that vision impairment and eye disease cost the US an estimated $68 billion annually in healthcare expenditures, reduced productivity, and diminished quality of life, with AMD itself having at least a $30 billion dollar negative impact on gross domestic product.

Diabetes is the leading cause of blindness among working-age adults in the United States. According to recent studies funded by the National Eye Institute, diabetic retinopathy, one of the most common and debilitating complications of diabetes, increased by 3.7 million new cases over the last decade. Approximately 7.7 million Americans are now affected by diabetic retinopathy. Even more alarming, the rate is projected to climb to 11 million by 2030. People with diabetes are also at greater risk for cataracts and glaucoma. But diabetic retinopathy (DR) is by far the most common sight-threatening condition among people with diabetes and is the leading cause of blindness in adults aged 20 to 74 years. Diabetic retinopathy has an enormous impact on national health care spending: Twenty-one percent of national medical expenditures for ophthalmic complications are attributable to diabetes.

The current standard of care for DR is to identify and treat the disease just before irreversible visual loss occurs. In practice, this means that accurate, early diagnosis of severe Non-Proliferative DR and/or Diabetic Macular Edema (DME) is needed to identify suitable candidates for Laser Photocoagulation, vitrectomy or Intra-vitreal Triamcinolone, as appropriate. Because DR is frequently asymptomatic, and any degree of DR is a risk factor for further progression, annual comprehensive eye exams are recommended for all individuals with diabetes.

Use of home - based smartphone visual acuity testing apps has the potential to diagnose and monitor the progression of DR at a very early stage of the disease and to monitor visual changes in macular degeneration. Additionally, The AREDS2-HOME study showed early detection of neovascular AMD resulted in better vision outcomes compared to standard monitoring of neovascular AMD. Identification of changes in vision would trigger further clinical attention and possible interventions. It is conceivable that this would ultimately reduce the economic burden of DR and AMD.

DigiSight's Checkup Vision Assessment System allows subjects to frequently check their vision in a rapid, quantitative and reproducible way, and transmit that information in a secure and organized fashion, enabling their physicians to optimize and administer treatment in a timely manner. We designed the CLEAR study to evaluate the agreement between Checkup Vision Assessment System and standard office based visual acuity tests. Because the Checkup test is a near vision test we are using the Lebensohn Near Card as the main comparator.

CLEAR STUDY OBJECTIVES:

* Evaluate the agreement of the Checkup Vision Assessment System (Checkup) with the reference device for assessing near visual acuity
* Evaluate the agreement of the Checkup Vision Assessment System (Checkup) with the reference device for assessing metamorphopsia .

OVERVIEW The CLEAR study is a prospective, single arm evaluation of the Paxos Checkup app tests, to be conducted in two phases under a common protocol. In the first phase the comparative performance of Checkup to the pre-specified reference methods in assessing near vision and in the presence of normal, AMD or DR was documented in 27 enrolled subjects. Results of the first phase were used to finalize the protocol and estimated sample size for Phase 2. There will be no formal statistical tests of Phase 1 results, and data from Phase 1 will not be pooled with Phase 2 results. The study will transition from Phase 1 to Phase 2 when it is believed that sufficient data have been collected in Phase 1 to plan and implement Phase 2 (pivotal). Phase 2 is planned to enroll 110 patients, based on evaluation of Phase I (pilot) results.

Subjects will be enrolled into three subpopulations based on eye health status: subjects with AMD (approximately 50% of total), subjects with DR (approximately 30% of total), and subjects with normal eye health (approximately 20% of total).

In Phase 2 the hypotheses associated with the two primary endpoints for the study will be statistically tested against pre-specified performance goals. These performance goals are based on the test-retest correlation of findings from the reference test methods in the study population.

Primary Endpoint 1:

Corrected Near Visual Acuity (CNVA) assessed with the Checkup System will be compared to the reference method CNVA (Lebensohn Near Card) in replicated measurements at each of two in-office visits.

Primary Endpoint 2:

The Amsler Grid assessment with the Checkup will be compared to the reference method Amsler Grid in replicated measurements at each of two in-office visits.

ELIGIBILITY:
Inclusion Criteria:

* Male or female 18 years of age and older
* Best Corrected Near Visual acuity 20/200 or better in study eye(s)
* Able and willing to make the required study visits
* Able and willing to provide consent and comply with study assessments for the full duration of the study.

Specific Inclusion Criteria for Subgroup with Normal Eyes

* Best Corrected Near Visual acuity 20/32 or better in each eye
* No concurrent systemic illness affecting the retina and vision.

Specific Inclusion Criteria for Subgroups with AMD or DR

* Diagnosis of either AMD or DR (all subgroups qualify)

Exclusion Criteria:

* Dementia or other neurologic or psychological limitation that would prevent the patient from performing regular self-testing of visual function
* Other comorbid ocular pathology affecting vision (with the exception of cataract, pseudophakia, refractive error, and/or presbyopia)
* Inability to successfully undergo training and certify ability to self-test with Paxos Checkup
* Inability to return for follow up

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Study population includes patients with no pathology, patients with Diabetic Retinopathy and patients with Adult Macular Degeneration.
Sampling Method: Non-Probability Sample
Enrollment: 143 (Actual)
Dates: Start 2016-07 (Actual); Primary Completion 2018-03 (Estimated); Study Completion 2018-03 (Estimated)

PRIMARY OUTCOMES:
Near Corrected Visual Acuity | Eight weeks
  Corrected Near Visual Acuity (CNVA) assessed with the Checkup System will be compared to the reference method CNVA (Lebensohn Near Card) in replicated measurements at each of two in-office visits.
Amsler Grid | Eight weeks
  The Amsler Grid assessment with the Checkup will be compared to the reference method Amsler Grid in replicated measurements at each of two in-office visits

SECONDARY OUTCOMES:
Feasibility of home testing using Paxos Checkup Mobile application | Eight weeks
  Assessment of study subjects ability to successfully complete a home test using the Feasibility of home testing measured by Paxos Checkup Mobile application.
Assess repeatability of mobile application testing | 8 weeks
  Assess the repeatability of in-office Checkup visual acuity and Amsler testing.

CONTACTS AND LOCATIONS:
Overall Officials: Carol Hoang, Study Director — Digisight Technologies, Inc.
Locations (12):
- United States (12):
  - Phoenix, Arizona
  - Mountain View, California
  - Fort Myers, Florida
  - Miami, Florida
  - Tallahassee, Florida
  - Lexington, Kentucky
  - Reno, Nevada
  - Cleveland, Ohio
  - Nashville, Tennessee
  - Austin, Texas
  - San Antonio, Texas
  - Spokane, Washington

IPD SHARING:
Plan to Share IPD: Undecided